CLINICAL TRIAL: NCT00399997
Title: Effect of Exercise on Prescription on Physical Activity, Physical Fitness, and Health in Patients With Lifestyle Diseases
Brief Title: Evaluation of Effect of Exercise on Prescription
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: The County of Vejle (Unknown); The County of Ribe (Unknown); The Danish Medical Research Council (Other); Ministry of the Interior and Health, Denmark (Other Government); National Board of Health, Denmark (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-04-0084 JBS
Record Dates: First submitted 2006-11-15; First posted 2006-11-16 (Estimated); Last update posted 2006-12-22 (Estimated); Status verified 2006-11

CONDITIONS: Metabolic Syndrome X; Diabetes Mellitus, Type 2; Cardiovascular Diseases
Keywords: Exercise; Exercise referral; Lifestyle diseases; Sedentary behavior
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus, Type 2; Cardiovascular Diseases; Motor Activity; Sedentary Behavior

INTERVENTIONS:
Behavioral: Exercise on Prescription

SUMMARY:
The purpose of this study is to evaluate the effect of a primary healthcare intervention called 'Exercise on Prescription' aimed at increasing level of physical activity in a population of sedentary patients with increased risk of developing lifestyle diseases. The effect is evaluated using both objective and patient-reported variables.

DETAILED DESCRIPTION:
Exercise prescriptions are used for initiating a physical active lifestyle in sedentary populations.

A Danish project called 'Exercise on Prescription' (EoP) is implemented in primary healthcare. Patients eligible for EoP are non-institutionalised adults with medically controlled lifestyle diseases or risk factors of lifestyle diseases, who are motivated to change lifestyle, able to improve health status through a physical active lifestyle, and willing to pay a fee of €100 for the intervention.

The purpose of this study is to assess the effect on: 1) maximal oxygen uptake (VO2max), 2) bodyweight and Body Mass Index, 3) glycemic control (in patients with impaired glucose tolerance), 4) physical activity level, and 5) health related quality of life.

The EoP-group is compared to a control group.

ELIGIBILITY:
Inclusion Criteria:

* all patients referred to the Exercise on Prescription scheme by their general practitioner
* volunteer to participate in the randomized trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-01; Study Completion 2007-08

PRIMARY OUTCOMES:
Maximal oxygen uptake at 4 and 10 months
Bodyweight and Body Mass Index at 4 and 10 months
Glycemic control at 4 and 10 months
Patient-reported physical activity level at 4 and 10 months
Patient-reported health related quality of life at 4 and 10 months

SECONDARY OUTCOMES:
Patient-reported amount and intensity of exercise at 4 and 10 months
Patient-reported physical fitness at 4 and 10 months
Patient-reported compliance with national guidelines for physical activity at 4 and 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Jes Bak Sørensen, MSc, Principal Investigator — Centre of Applied and Clinical Exercise Sciences, Institute of Sports Science and Clinical Biomechanics, University of Southern Denmark
Locations (1):
- Centre of Applied and Clinical Exercise Sciences, Institute of Sports Science and Clinical Biomechanics, University of Southern Denmark, Odense, Denmark

REFERENCES:
- [Background] Sorensen JB, Skovgaard T, Puggaard L. Exercise on prescription in general practice: a systematic review. Scand J Prim Health Care. 2006 Jun;24(2):69-74. doi: 10.1080/02813430600700027. PMID 16690553